CLINICAL TRIAL: NCT06073002
Title: Effects of a Home-Based Exercise Intervention on Physical Function, Symptoms and Health-Related Quality of Life in Subjects with Long Covid
Brief Title: Effects of a Home-Based Exercise Intervention in Subjects with Long COVID
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Daniel König, Principal Investigator, University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 01017
Record Dates: First submitted 2023-10-06; First posted 2023-10-10 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Long COVID-19; Post-COVID-19 Syndrome
Keywords: exercise; exercise therapy; concurrent training; exercise rehabilitation; Long COVID-19; Post-COVID-19 Syndrome; home-based training
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Home-based concurrent training (Experimental): Combination of resistance training (5 exercises with bodyweight and/or resistance bands; 3 sets per exercise, 15-20 repetitions) and endurance training (mode of choice, light to moderate intensities which are monitored via heartrate zones, 20-40min per sessions); 3 weekly sessions on non-consecutive days
  Interventions: Other: home-based concurrent exercise

INTERVENTIONS:
Other: home-based concurrent exercise — 3 weekly sessions of home-based concurrent exercise on non-consecutive days. Resistance exercise is comprised of lunges, hip thrusts, pushups, resistance band rows, core and performed for 3 sets with 15-20 repetitions at an RPE of 14-18 (6-20 BORG scale). Endurance exercise can be done by the mode of choice and is monitored by heartrate zones. Sessions are of low to moderate intensity (below VT2) and the duration will be slowly increased for 20-40min.

SUMMARY:
The current Coronavirus Disease 2019 (COVID-19) pandemic is the most severe health crisis of the 21st century. This is not only due to the deaths caused by the disease. People that were affected by COVID-19 and supposedly recovered may suffer from long lasting sequelae. The presence of symptoms longer than 3 months after the infection with the Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) is referred to as Post-COVID-19 Syndrome or Long COVID-19. It is estimated that 10-20 percent of all infected people are affected. The most common symptoms include persistent fatigue, reduced physical capacity, dyspnoea, ageusia, anosmia, musculoskeletal pain and neuropsychological complaints such as depression, anxiety, insomnia and a loss of concentration.

Considering the novelty of the pathology, evidence on the successful treatment of Post-COVID/Long-COVID is scarce. Physical activity has been established as a treatment option for chronic diseases that have similar symptomatic manifestations to those of Post-COVID/Long-COVID. For example, exercise therapy has shown positive effects on the health status of patients with lung disease, depression, anxiety, insomnia and cognitive impairment. However, there has been controversy whether so-called Graded Exercise Therapy (GET) is a safe treatment strategy for patients with Chronic Fatigue Syndrome (CFS). This population may experience Post Exertional Malaise (PEM), a worsening of symptoms after physical, cognitive or emotional exertion. Since COVID-19 might be an infectious trigger for CFS, particular caution has to be taken when recruiting participants and when screening them for adverse events and worsening of symptoms during an exercise intervention.

It can be hypothesized that patients suffering from Post-COVID/Long-COVID can benefit from exercise in various ways, guaranteed that there is sufficient screening for PEM before and during the intervention and training volume and intensity are increased slowly and progressively.

The current study investigates the effects of a home-based concurrent training program on various parameters in people affected by Long COVID.

ELIGIBILITY:
Inclusion Criteria:

* laboratory-confirmed infection with SARS-CoV-2 via PCR a minimum of 12 weeks ago
* presence of at least one or more of persistent symptoms that can be attributed to Long-COVID

Exclusion Criteria:

* previous or current hospitalization due to the COVID-19 disease
* regular engagement in endurance or strength training (more than once per week) in the six months prior to enrollment
* contraindications for physical endurance and resistance exercise according to the guidelines of the American College of Sports Medicine (ACSM)
* a grade of 3 or higher on the Post-COVID-19 Functional Status Scale (PCFS)
* presence of post exertional malaise (PEM)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Change of peak oxygen consumption (VO2peak measured in ml/min/kg) | at baseline and at 12 weeks
  VO2peak will be assessed during cardio pulmonary exercise testing (CPET) on a bicycle ergometer.

SECONDARY OUTCOMES:
Change of maximum lower body isometric muscle strength (measured in N) | at baseline and at 12 weeks
  Maximum lower body isometric muscle strength will be assessed via a leg press with integrated isometric force measurement (Compass 530, Suessmed GmbH).
Change of maximum hand grip strength (measured in kg) | at baseline and at 12 weeks
  Maximum hand grip strength will be assessed via a hand grip dynamometer (Saehan SH5001).
Change of Standard Deviation of RR-Intervals (SDNN measured in ms) | at baseline and at 12 weeks
  SDNN will be assessed via a short-term heart rate variability (HRV) measurement (BioSign).
Change of Root Mean Square of Successive Differences (RMSSD measured in ms) | at baseline and at 12 weeks
  RMSSD will be assessed via a short-term heart rate variability (HRV) measurement (BioSign).
Change of health-related quality of life (HQoL) assessed via the SF-36 1.0 | at baseline an at 12 weeks
  The SF-36 1.0 is self-administered questionnaire and will be scored according to RAND (numeric value of 0-100). A high score represents a more favorable health status.
Change of the number of present Long-COVID specific symptoms | at baseline and at 12 weeks
  The number of Long-COVID specific symptoms will be assessed using a list of symptoms provided by the National Institute for Health Care and Excellence (NICE). Each item will be referenced to as existent (yes) or non-existent (no) during the last 7 days.
Change of fatigue assessed via the Fatigue Severity Scale (FSS) | at baseline and at 12 weeks
  The FSS is a 9-item self-report questionnaire using a 1-7 Likert-scale
Change of dyspnoea assessed via the modified Medical Research Council (mMRC) dyspnoea scale | at baseline and at 12 weeks
  The mMRC dyspnoea scale measures perceived breathlessness and classifies subjects into dyspnoea grades from 0-4.
Change of interleukin-6 (IL-6 measured in pg/ml) | at baseline and at 12 weeks
  IL-6 will be assessed via blood sample.
Change of tumor necrosis factor alpha (TNF-α measured in pg/ml) | at baseline and at 12 weeks
  TNF-α will be assessed via blood sample.
Change of mean time "correct rejection" (CR, speed during concentrated working measured in s) | at baseline and at 12 weeks
  CR will be assessed via Cognitrone (Schuhfried GmbH), which is a carefully administered computer test. Participants will be given the task of comparing a series of geometric figures.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sport and Human Movement Science, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No